CLINICAL TRIAL: NCT04567368
Title: Two-site Laboratory-based Diagnostic Accuracy and Feasibility Study of the Xpert MTB/XDR Assay for Detection of Isoniazid, Fluoroquinolone, Ethionamide and Second-line Injectable Anti-tuberculosis Drug Resistance
Brief Title: TB-CAPT MTB/XDR Study
Status: Active, not recruiting | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: University of Cape Town (Other); Wits Health Consortium (Pty) Ltd (Other); Ludwig-Maximilians - University of Munich (Other); Ospedale San Raffaele (Other); Swiss Tropical & Public Health Institute (Other); Heidelberg University (Other); African Society for Laboratory Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: TB042
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Tuberculosis; Resistance Bacterial; Diagnoses Disease
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Xpert MTB/XDR — Cepheid Xpert MTB/XDR assay for detection of resistance to INH, FQ and SLID

SUMMARY:
The Cepheid Xpert MTB/XDR cartridge, which runs on the same platform as Xpert MTB/RIF Ultra, has been developed to detect additional resistance to isoniazid, fluoroquinolones and second-line injectable anti-tuberculosis drugs and provides results within 2 hours and on primary samples. An evaluation of the the Xpert MTB/XDR assay is currently underway in clinical settings in South Africa, India and Moldova. The TB-CAPT MTB/XDR Study will add further diagnostic accuracy and feasibility data to the evidence base for the Xpert MTB/XDR assay.

ELIGIBILITY:
Inclusion Criteria:

* Mtb-positive, rifampicin-resistant respiratory specimen identified on Xpert MTB/RIF Ultra

Exclusion Criteria:

* Residual SR-sputum mix not retained or not found
* Patient previously included in the study

Exclusion for diagnostic accuracy and time-to-result endpoints:

* Insufficient residual SR-sputum mix remaining for Xpert MTB/XDR (<2 ml)
* Xpert MTB/XDR unsuccessful
* No second / follow-up specimen received
* Second / follow-up specimen culture-negative, contaminated or not available
* Reference standard uninterpretable (phenotyping or WGS)

  * Where phenotypic susceptibility testing results are uninterpretable, specimens will still be included in WGS comparison
  * Where WGS results are uninterpretable, specimens will still be included in phenotypic susceptibility testing comparison

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Respiratory specimens testing rifampicin-resistant Mtb positive on Xpert MTB/RIF Ultra.
  The proposed study procedures would not affect the usual care of patients as we will utilise specimens that would ordinarily be discarded. Similarly, the reference standard tests (next generation sequencing) are non-routine tests not currently utilised for patient care in South Africa. These tests will be performed post hoc with patient identifiers removed.
  For these reasons, we are proposing a waiver of informed consent for this diagnostic accuracy and feasibility study.
Sampling Method: Non-Probability Sample
Enrollment: 753 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of Xpert MTB/XDR assay | enrolment
  Sensitivity and specificity of Xpert MTB/XDR assay vs. the composite reference standard for detection of resistance to Isoniazid, Fluoroquinolones, Ethionamide, Second-line injectable anti-tuberculosis drugs

SECONDARY OUTCOMES:
Sensitivity and specificity of Xpert MTB/XDR assay compared to phenotypic anti-tuberculosis drug susceptibility testing and WGS separately | enrolment
  Sensitivity and specificity of Xpert MTB/XDR assay for detection of resistance to Isoniazid, Fluoroquinolones, Ethionamide, Second-line injectable anti-tuberculosis drugs compared to phenotypic anti-tuberculosis drug susceptibility testing and WGS separately

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - University of Cape Town, Cape Town
  - University of the Witwatersrand, Johannesburg

DOCUMENTS (2):
  • Study Protocol (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT04567368/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT04567368/SAP_001.pdf